CLINICAL TRIAL: NCT07127380
Title: MID-MIS Trail Protocol - Comparison of Clinical Outcomes, Complications Rate and Treatment Costs of Mini-TLIF and MIDLIF in the Treatment of Discogenic Low Back Pain
Brief Title: Comparison of Clinical Outcomes, Complications Rate and Treatment Costs of Mini-TLIF and MIDLIF in the Treatment of Discogenic Low Back Pain
Acronym: MID-MIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copernicus Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kamil Krystkiewicz, MD, PhD, neurosurgeon, Copernicus Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112/2024
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Lower Back Pain Chronic; Lumbar Degenerative Disease; Lumbar Disc Degeneration; Degenerative Disc Disease(DDD)
Keywords: Degenerative Disc Disease; Lower Back Pain; Lumbar Disc Degeneration; Discogenic Pain; MIS-TLIF; MIDLIF; mini-TLIF; Minimally Invasive Transforaminal Lumbar Interbody Fusion; Midline Lumbar Interbody Fusion; Spinal stabilization; Spinal fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Transforaminal Lumbar Interbody Fusion (mini-TLIF) (Active Comparator): Lumbar fusion is obatained by Minimally Invasive Transforaminal Lumbar Interbody Fusion
  Interventions: Procedure: Minimally Invasive Transforaminal Lumbar Interbody Fusion (mini-TLIF)
- Midline Lumbar Interbody Fusion (MIDLIF) (Experimental): Lumbar fusion is obtained by Midline Lumbar Interbody Fusion
  Interventions: Procedure: Midline Lumbar Interbody Fusion (MIDLIF)

INTERVENTIONS:
Procedure: Midline Lumbar Interbody Fusion (MIDLIF) — Midline Lumbar Interbody Fusion (MIDLIF) is a procedure utilizes a medial approach to the spine, involving the retraction of the segmental back muscles to expose the lamine and articular processes. Screw placement is medialized, with entry to a point along the pars intercularis or joint surface. It places the screw through potentially more cortical and stronger bone. Decompression is achieved by resecting the inferior articular process and lamina marginalis, followed by a discectomy. Subsequently, a transforaminal lumbar interbody fusion (TLIF) is performed to place an interbody cage and promote fusion.
  Arms: Midline Lumbar Interbody Fusion (MIDLIF)
Procedure: Minimally Invasive Transforaminal Lumbar Interbody Fusion (mini-TLIF) — Minimally invasive Transforaminal Lumbar Interbody Fusion (mini-TLIF) is a procedure that employs a percutaneous approach for pedicle screw placement through the pedicles. Decompression is performed using a lateral approach, with 2-3 cm lateral to the ipsilateral borders. This is followed by resection of the inferior articular process and removal of the ligamentum flavum, facilitating discectomy. An interbody cage is then inserted to achieve fusion.
  Arms: Minimally Invasive Transforaminal Lumbar Interbody Fusion (mini-TLIF)

SUMMARY:
Background

Degenerative disc disease (DDD) is the leading cause of lower back pain and disability, which prevalence increasing with age. When conservative treatment fails, surgical methods of spinal fusion are employed. Minimally invasive techniques, including minimally invasive transforaminal lumbar interbody fusion (MIS-TLIF) and midline lumbar interbody fusion (MIDLIF), have well-documented advantages over traditional open transforaminal interbody fusion (open-TLIF). However, data comparing these two minimally invasive methods in treating DDD are minimal and sometimes contradictory. I am running a few minutes late; my previous meeting is running over.

Methods This is a prospective, randomized, partially blinded, two-arm trial aiming to compare the outcomes, complications, and treatment costs of MIS-TLIF and MIDLIF in patients with discogenic low back pain. A total of 100 adult patients with lumbosacral spine pain and radicular symptoms, unresponsive to conservative treatment for over one year, will be enrolled. Patients will be randomized (1:1) into two arms: MIS-TLIF (control, n=50) and MIDLIF (intervention, n=50), with a 12-month follow-up. Inclusion criteria include age ≥18 years and discopathy at one or two levels requiring interbody stabilization. Exclusion criteria include multilevel pathology, spinal deformities, and pain causes other than degenerative disease. Primary endpoints assess pain (VAS, NRS scales), disability (COMI, ODI questionnaires), and quality of life (EQ-5D-5L questionnaire) at 1, 3, 6, and 12 months post-surgery. Secondary endpoints include complication rates (nerve root damage, infections), costs (hospitalization, implants), length of hospital stay, procedure duration, blood loss, morphometric parameters (intervertebral space height), and adjacent segment disease based on imaging studies (MRI, CT, X-ray). Data analysis uses parametric/non-parametric tests (e.g., t-test, Mann-Whitney) in the R software. The trial adheres to the Helsinki Declaration, with ethics approval (no. 112/2024).

Discussion Data on the comparison of MIDLIF and MIS-TLIF in treating DDD are minimal and inconsistent. Some reports have advantaged MIDLIF in shorter operative time, decreased intraoperative blood loss, and reduced hospital stays, while others favor MIS-TLIF. This trial addresses these gaps by providing high-quality evidence on clinical superiority, cost-effectiveness, and long-term outcomes compering MIDLIF and MIS-TLIF. There is a high need for a high-quality, prospective study to examine this problem.

ELIGIBILITY:
Inclusion Criteria:

* Discogenic lower lumbar-sacral pain lasting longer than one year
* Failure of conservative treatment, including rehabilitation and pain management
* Lumbar discopathy qualified for interbody fusion and pedicle screw stabilization
* Informed consent of the patient for the study and proposed treatment

Exclusion Criteria:

* Contraindications to surgery under general anesthesia
* Age < 18 years
* Pregnancy, breastfeeding
* Lack of informed consent to participate in the study
* Lumbar-sac discopathy requiring surgical treatment at more than two levels
* Spinal deformities: adult idiopathic scoliosis, degenerative scoliosis, deformity due to spinal malignancy, inflammatory spinal disease, post-traumatic, or associated with congenital anomalies
* Lower lumbar-sacral pain syndrome, which, in the investigator's opinion, has an etiology other than degenerative spine disease (e.g., cancer-related pain, ankylosing spondylitis)
* Spinal oncology disease
* True and degenerative spondylolisthesis
* Contraindications to performing MRI of the lumbar-sacral spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 1 day before randomization, up to 24 hours after randomization, 2 days after randomization, 1 month after randomization, 3 months after randomization, 6 months after randomization, 12 months after randomization
  The Visual Analog Scale (VAS) is a measurement tool designed to quantify subjective pain intensity. It consists of a straight horizontal line, typically 10 cm (100 mm) long, with two endpoints anchored by descriptive labels ("no pain" on the left and "worst imaginable pain" on the right). Respondents mark a point on the line that best represents their perception, and the score is determined by measuring the distance in millimeters from the left endpoint to the mark, yielding a continuous score from 0 to 100.
Numeric Rating Scale (NRS) | 1 day before randomization, up to 24 hours after randomization, 2 days after randomization, 1 month after randomization, 3 months after randomization, 6 months after randomization, 12 months after randomization
  The Numeric Rating Scale (NRS) is a unidimensional, self-reported psychometric tool primarily used to quantify the intensity of pain on a numerical scale. It typically consists of an 11-point scale ranging from 0 to 10, where 0 represents "no pain" (or no symptom) and 10 represents "worst possible pain" (or maximum intensity imaginable). Respondents verbally or in writing select a whole number that best reflects their current experience, making it a discrete rather than continuous measure.
Core Outcome Measures Index | 1 day before randomization, up to 24 hours after randomization, 2 days after randomization, 1 month after randomization, 3 months after randomization, 6 months after randomization, 12 months after randomization
  The Core Outcome Measures Index (COMI) is a multidimensional, patient-reported outcome measure designed to assess the key domains affected by spinal disorders, particularly low back pain and related conditions. It consists of a brief questionnaire (typically 7-8 items) that evaluates pain intensity, function, symptom-specific well-being, general quality of life, and disability (both social and work-related). Responses are scored on a 0-10 scale, where higher scores indicate worse outcomes; the overall COMI score is the average of the domain scores, providing a single summary index.
Oswestry Disability Index (ODI) | 1 day before randomization, up to 24 hours after randomization, 2 days after randomization, 1 month after randomization, 3 months after randomization, 6 months after randomization, 12 months after randomization
  The Oswestry Disability Index (ODI) is a self-reported questionnaire designed to quantify the level of functional disability associated with low back pain and related spinal conditions. It consists of 10 sections, each addressing a specific aspect of daily life impacted by pain: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life (optional in some versions), social life, and traveling. Each section has 6 statements scored from 0 (no limitation) to 5 (maximum limitation), with the total score expressed as a percentage (0-100%), where higher scores indicate greater disability. Common interpretations include 0-20% (minimal disability), 21-40% (moderate), 41-60% (severe), 61-80% (crippled), and 81-100% (bed-bound or exaggerating symptoms).
European Quality of Life - 5 Dimensions, 5 Levels | 1 day before randomization, up to 24 hours after randomization, 2 days after randomization, 1 month after randomization, 3 months after randomization, 6 months after randomization, 12 months after randomization
  The European Quality of Life - 5 Dimensions, 5 Levels (EQ-5D-5L) is a standardized, self-reported instrument developed by the EuroQol Group to measure health-related quality of life (HRQoL) across a wide range of populations and conditions. It comprises two main components: a descriptive system with five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels of severity.

SECONDARY OUTCOMES:
Complication Rates and Types | Up to 24 hours after randomization, 2 days after randomization, 1 month after randomization, 3 months after randomization, 6 months after randomization, 12 months after randomization
  Evaluation of the frequency and nature of complications between groups, including nerve root damage, cerebrospinal fluid leak, instrumentation failure, postoperative wound infection, and other adverse events.
Direct Treatment Costs | 12 months after randomization
  Analysis of direct treatment costs with a breakdown by category, including total hospitalization costs, costs of implants used, costs of medications administered, and costs of the surgical procedure.
Hospitalization Duration | 2 days after randomization (day of hospital discharge)
  Measurement of the length of stay (LOS) in the hospital.
Procedure Duration | 2 days after randomization
  Evaluation of the operating room time (OR time) required for the surgery.
Blood Loss | 2 days after randomization
  Quantification of estimated blood loss (EBL) during the surgical procedure.
Spinal Morphometric Parameters | 2 days after randomization, 3 months after randomization, 12 months after randomization
  Evaluation of intervertebral space height (ISH), foraminal height (FH), radiological evidence of bone fusion, and global and segmental lordosis of the lumbar-sacral spine.
Time to Return to Professional Activity | 12 months after randomization
  Measurement of the duration required for working patients to resume professional activities.
Radiological Assessment of Adjacent Segment Disease | 12 months after randomization
  Evaluation of the occurrence of adjacent segment disease based on MRI of the lumbar-sacral spine.

CONTACTS AND LOCATIONS:
Locations (1):
- Copernicus Memorial Hospital in Łódź, Poland, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva PS, Jardim A, Pereira J, Sousa R, Vaz R, Pereira P. Minimally invasive fusion surgery for patients with degenerative spondylolisthesis and severe lumbar spinal stenosis: a comparative study between MIDLIF and TLIF. Eur Spine J. 2023 Sep;32(9):3210-3217. doi: 10.1007/s00586-023-07847-6. Epub 2023 Jul 9. PMID 37422769
- [Background] Tippins NP, Foreit AM, Kussow NJ, Milne CM, Narayanan AM, Neely MR, Poplarski JH, Reasoner JT, Ricks K, Alentado VJ, Potts EA, Mobasser JP. Examination of clinical and radiographic outcomes after lumbar interbody fusion: a retrospective analysis of TLIF, MidLIF, and MIS-TLIF procedures. J Neurosurg Spine. 2025 May 2;43(1):52-62. doi: 10.3171/2025.1.SPINE241286. Print 2025 Jul 1. PMID 40315609
- [Background] Crawford CH 3rd, Owens RK 2nd, Djurasovic M, Gum JL, Dimar JR 2nd, Carreon LY. Minimally-Invasive midline posterior interbody fusion with cortical bone trajectory screws compares favorably to traditional open transforaminal interbody fusion. Heliyon. 2019 Sep 11;5(9):e02423. doi: 10.1016/j.heliyon.2019.e02423. eCollection 2019 Sep. PMID 31535047
- [Background] Parker SL, Adogwa O, Witham TF, Aaronson OS, Cheng J, McGirt MJ. Post-operative infection after minimally invasive versus open transforaminal lumbar interbody fusion (TLIF): literature review and cost analysis. Minim Invasive Neurosurg. 2011 Feb;54(1):33-7. doi: 10.1055/s-0030-1269904. Epub 2011 Apr 19. PMID 21506066
- [Background] Xie L, Wu WJ, Liang Y. Comparison between Minimally Invasive Transforaminal Lumbar Interbody Fusion and Conventional Open Transforaminal Lumbar Interbody Fusion: An Updated Meta-analysis. Chin Med J (Engl). 2016 Aug 20;129(16):1969-86. doi: 10.4103/0366-6999.187847. PMID 27503024
- [Background] Xue J, Song Y, Liu H, Liu L, Li T, Gong Q. Minimally invasive versus open transforaminal lumbar interbody fusion for single segmental lumbar disc herniation: A meta-analysis. J Back Musculoskelet Rehabil. 2022;35(3):505-516. doi: 10.3233/BMR-210004. PMID 34602458
- [Background] Heemskerk JL, Oluwadara Akinduro O, Clifton W, Quinones-Hinojosa A, Abode-Iyamah KO. Long-term clinical outcome of minimally invasive versus open single-level transforaminal lumbar interbody fusion for degenerative lumbar diseases: a meta-analysis. Spine J. 2021 Dec;21(12):2049-2065. doi: 10.1016/j.spinee.2021.07.006. Epub 2021 Jul 14. PMID 34273567
- [Background] Phani Kiran S, Sudhir G. Minimally invasive transforaminal lumbar interbody fusion - A narrative review on the present status. J Clin Orthop Trauma. 2021 Sep 8;22:101592. doi: 10.1016/j.jcot.2021.101592. eCollection 2021 Nov. PMID 34603954
- [Background] Zhang X, Zhang Y, Gu Z, Li G. Comparison of midline lumbar interbody fusion and minimally invasive transforaminal lumbar interbody fusion for treatment of lumbar degeneration disease. Sci Rep. 2024 Sep 27;14(1):22154. doi: 10.1038/s41598-024-73213-1. PMID 39333680
- [Background] Wang YY, Chung YH, Huang CH, Hu MH. Comparison of minimally invasive transforaminal lumbar interbody fusion and midline lumbar interbody fusion in patients with spondylolisthesis. J Orthop Surg Res. 2024 May 9;19(1):286. doi: 10.1186/s13018-024-04764-2. PMID 38725087
- [Background] Silva F, Silva PS, Vaz R, Pereira P. Midline lumbar interbody fusion (MIDLIF) with cortical screws: initial experience and learning curve. Acta Neurochir (Wien). 2019 Dec;161(12):2415-2420. doi: 10.1007/s00701-019-04079-w. Epub 2019 Oct 24. PMID 31650331
- [Background] Dave BR, Marathe N, Mayi S, Degulmadi D, Rai RR, Patil S, Jadav K, Bali SK, Kumar A, Meena U, Parmar V, Amin P, Dave M, Krishnan PA, Krishnan A. Does Conventional Open TLIF cause more Muscle Injury when Compared to Minimally Invasive TLIF?-A Prospective Single Center Analysis. Global Spine J. 2024 Jan;14(1):93-100. doi: 10.1177/21925682221095467. Epub 2022 Apr 20. PMID 35442112
- [Background] Modi HN, Shrestha U. Comparison of Clinical Outcome and Radiologic Parameters in Open TLIF Versus MIS-TLIF in Single- or Double-Level Lumbar Surgeries. Int J Spine Surg. 2021 Oct;15(5):962-970. doi: 10.14444/8126. Epub 2021 Sep 22. PMID 34551928
- [Background] Tan JH, Liu G, Ng R, Kumar N, Wong HK, Liu G. Is MIS-TLIF superior to open TLIF in obese patients?: A systematic review and meta-analysis. Eur Spine J. 2018 Aug;27(8):1877-1886. doi: 10.1007/s00586-018-5630-0. Epub 2018 Jun 1. PMID 29858673
- [Background] Mobbs RJ, Phan K, Malham G, Seex K, Rao PJ. Lumbar interbody fusion: techniques, indications and comparison of interbody fusion options including PLIF, TLIF, MI-TLIF, OLIF/ATP, LLIF and ALIF. J Spine Surg. 2015 Dec;1(1):2-18. doi: 10.3978/j.issn.2414-469X.2015.10.05. PMID 27683674
- [Background] Mohd Isa IL, Teoh SL, Mohd Nor NH, Mokhtar SA. Discogenic Low Back Pain: Anatomy, Pathophysiology and Treatments of Intervertebral Disc Degeneration. Int J Mol Sci. 2022 Dec 22;24(1):208. doi: 10.3390/ijms24010208. PMID 36613651
- [Background] Wu PH, Kim HS, Jang IT. Intervertebral Disc Diseases PART 2: A Review of the Current Diagnostic and Treatment Strategies for Intervertebral Disc Disease. Int J Mol Sci. 2020 Mar 20;21(6):2135. doi: 10.3390/ijms21062135. PMID 32244936
- [Background] Chou R. Low Back Pain. Ann Intern Med. 2021 Aug;174(8):ITC113-ITC128. doi: 10.7326/AITC202108170. Epub 2021 Aug 10. PMID 34370518